CLINICAL TRIAL: NCT06630130
Title: A Phase II Platform Trial of Perioperative Therapies in Locally Advanced Unresectable Gastric Cancer (Neo-VIKTORY)
Brief Title: Perioperative Therapies in Locally Advanced Unresectable Gastric Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jeeyun Lee (Other)
Responsible Party: Sponsor-Investigator, Jeeyun Lee, Professor, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-07-077
Record Dates: First submitted 2024-08-01; First posted 2024-10-08 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms | interventions — trastuzumab deruxtecan; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A : T-DXd and Capecitabine combination (Active Comparator): Neoadjuvant; Trastuzumab Deruxtecan(T-DXd) 5.4mg/kg IV on D1 and Capecitabine 1000mg/m2 PO BID on D1-D14, Q3W for 3 cycles
  -Adjuvant; Trastuzumab Deruxtecan(T-DXd) 5.4mg/kg IV on D1, Q3W 16 cycles (up to 12 months) and Capecitabine 1000mg/m2 PO BID on D1-D14, Q3W for 4 cycles (up to 3 months)
  Interventions: Drug: Trastuzumab deruxtecan; Drug: Capecitabine
- Cohort B : T-DXd and Capecitabine and Rilvegostomig combination (Active Comparator): * Neoadjuvant; Trastuzumab Deruxtecan(T-DXd) 5.4mg/kg IV on D1 and Capecitabine 1000mg/m2 PO BID on D1-D14 with Rilvegostomig 750mg IV on D1, Q3W for 3 cycles
  * Adjuvant; Trastuzumab Deruxtecan(T-DXd) 5.4mg/kg IV with Rilvegostomig 750mg IV on D1, Q3W for 16 cycles (up to 12 months) and Capecitabine 1000mg/m2 PO BID on D1-D14, Q3W for 4 cycles (up to 3 months)
  Interventions: Drug: Trastuzumab deruxtecan; Drug: Capecitabine; Drug: Rilvegostomig

INTERVENTIONS:
Drug: Trastuzumab deruxtecan — * Neoadjuvant; Trastuzumab Deruxtecan(T-DXd) 5.4mg/kg IV on D1, Q3W for 3 cycles
  * Adjuvant; Trastuzumab Deruxtecan(T-DXd) 5.4mg/kg IV on D1, Q3W 16 cycles (up to 12 months)
  Other Names: Enhertu
Drug: Capecitabine — * Neoadjuvant; Capecitabine 1000mg/m2 PO BID on D1-D14, Q3W for 3 cycles
  * Adjuvant; Capecitabine 1000mg/m2 PO BID on D1-D14, Q3W for 4 cycles (up to 3 months)
  Other Names: Xeloda
Drug: Rilvegostomig — (Only Cohort B)
  * Neoadjuvant; Rilvegostomig 750mg IV on D1, Q3W for 3 cycles
  * Adjuvant; Rilvegostomig 750mg IV on D1, Q3W for 16 cycles (up to 12 months)
  Other Names: AZD2936
  Arms: Cohort B : T-DXd and Capecitabine and Rilvegostomig combination

SUMMARY:
Gastric cancer (GC) is the fifth most commonly diagnosed cancer, with over one million cases diagnosed annually worldwide. Human epidermal growth factor receptor 2 (HER2) overexpression in GC (seen in 4.4% to 53.4% of patients in different reports) is predictive biomarker of response to HER2-targeting therapies.

Trastuzumab in combination with cisplatin or oxaliplatin, and a fluoropyrimidine (capecitabine or 5-fluorouracil [5-FU]), is approved anti-HER2 therapy for first-line treatment of HER2-positive gastric or gastroesophageal junction (GEJ) cancer.

Rilvegostomig 750 mg Q3W was selected as recommended Phase 2 dose based on all available ARTEMIDE-01 clinical safety, efficacy, PK, RO data as well as modeling analysis. The dose of 750 mg Q3W is predicted to achieve intra-tumoral RO of ≥ 90% in the majority of participants across a broad spectrum of conditions.

This is a phase II study to initially assess the efficacy of perioperative Trastuzumab Deruxtecan (T-DXd) and Capecitabine combination with or without Rilvegostomig in patients with HER2 positive locally advanced unresectable GC and potentially by subsequent protocol amendment in HER2 low locally advanced GC. Other agents may also subsequently be assessed in this protocol, by protocol amendments

DETAILED DESCRIPTION:
Neoadjuvant therapy will begin following completion of the screening period, and patients will undergo resection surgery 4 to 8 weeks after the last dose of neoadjuvant therapy. Surgery >8 weeks after the last dose of neoadjuvant therapy may be permitted in consultation with the Sponsor. Adjuvant therapy will begin 4 to 12weeks post-surgery (based on the patient's recovery period).

Tumor evaluation using modified RECIST 1.1 will be conducted at screening (within 28 days prior to first dose) and ≤28 days after last dose of neoadjuvant therapy and after surgery.

Every 12 weeks (±1 week) relative to the Adjuvant Baseline scan for first years and then every 24 weeks (±2 week) until progression/recurrence

The imaging modalities used for modified RECIST 1.1 assessment will be CT or MRI scans of chest, abdomen and pelvis. Modified RECIST 1.1 scans will be analyzed by the investigator on site.

ELIGIBILITY:
Inclusion Criteria:

* 1. Provision of fully informed consent prior to any study specific procedures.
* 2. Patients must be ≥ 19 years of age
* 3. Body weight > 30kg
* 4. Has a Pathologically documented adenocarcinoma of gastric or gastroesophageal junction with HER2 IHC results.
* 5. In initial Cohort, HER2 positive (HER2 IHC 3+ or HER2 IHC 2+/ISH positive))
* 6. Locally advanced unresectable disease by physician's discretion (ex. cT4 or bulky Nx node or localized peritoneal seeding) No evident distant organ metastasis.
* 7. ECOG performance status PS 0-1 with no deterioration between screening and the first dose of study treatment.
* 8. Has LVEF ≥ 50% by either echocardiogram (ECHO) or multi-gated acquisition (MUGA) scan within 28 days before treatment
* 9. Has measurable target disease assessed by the Investigator based on RECIST version 1.1.
* 10. Has adequate organ and bone marrow, liver and renal function within 14 days before treatment (Note: Transfusion (red blood cell or platelet) or G-CSF administration is not allowed within 14 days prior to the day on which bone marrow function is assessed, or at any time after this day and prior to C1D1.)

  1. Hemoglobin ≥ 9.0 g/dL (≥8.0 g/dL in GC Indications)
  2. Platelet count ≥100 x 109/L
  3. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
  4. Total bilirubin ≤ 1.5 ULN if no liver metastases < 3×ULN in the presence of documented Gilbert's syndrome (unconjugated hyperbilirubinemia) or liver metastases at baseline
  5. AST (SGOT)/ALT (SGPT) ≤ 3.0 x ULN (< 5×ULN in participants with liver metastases)
  6. Serum albumin ≥ 2.5 g/dL
  7. CrCL(Ccr) ≥30mL/min (> 45ml/min in Rilvegostomig) as determined by Cockcroft Gault (using actual body weight)
  8. International normalized ratio or Prothrombin time and either partial thromboplastin or activated partial thromboplastin time ≤ 1.5 × ULN
* 11. Female patients must be using a highly effective method of contraception (refer to the restrictions on P45) during the clinical trial and for 7 months after permanent discontinuation of the study drug. There must be evidence that patients are not breastfeeding, have a negative pregnancy test, or not of childbearing potential by meeting one of the following criteria at screening:

  1. Post-menopausal women defined as aged more than 50 years and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatment.
  2. Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy, but not tubal ligation.
  3. Amenorrhoeic for 12 months and serum follicle-stimulating hormone (FSH), luteinizing hormone (LH) and plasma oestradiol levels in the postmenopausal range for the institution.

     More detailed information is provided in Appendix G (Definition and accepted contraception for women of childbearing age). Also female participants must not breastfeed and must not donate/retrieve ova from screening to 60days post last dose.
* 12. Non-sterilized male patients who are sexually active with a female partner of childbearing potential must use a condom with spermicide from screening to 4 months after the final dose of IMP. Complete heterosexual abstinence for the duration of the study and drug washout period is an acceptable contraceptive method if it is in line with the patient's usual lifestyle (consideration must be made to the duration of the clinical trial); however, periodic or occasional abstinence, the rhythm method, and the withdrawal method are not acceptable. It is strongly recommended for the female partners of a male patient to also use at least one highly effective method of contraception throughout this period. In addition, male patients should refrain from fathering a child, or freezing or donating sperm from the time of randomization/enrolment, throughout the study and for 4 months after the last dose of IMP. Preservation of sperm should be considered prior to enrollment in this study.

Exclusion Criteria:

* 1. Patients with evident peritoneal metastasis (including tumor cells in peritoneal fluid) or distant metastasis
* 2. Known dihydropyrimidine dehydrogenase (DPD) enzyme deficiency based on either local or central laboratory testing. Central laboratory testing will be available for patients where testing is SOC and with unknown DPD status.
* 3. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, uncontrolled hypertension, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs, or compromise the ability of the participant to give written informed consent.
* 4. Unresolved toxicities of ≥ Grade 2 (Common Terminology Criteria for Adverse Events [CTCAE] v5.0) from prior therapy (excluding vitiligo, alopecia, endocrine disorders that are controlled with replacement hormone therapy, asymptomatic laboratory abnormalities).
* 5. History of organ transplant.
* 6. Active primary immunodeficiency/active infectious diseases. Active or prior documented autoimmune or inflammatory disorders (including IBD [e.g. Crohn's disease, ulcerative colitis or diverticulitis], SLE, sarcoidosis syndrome, tuberculosis, Wegener syndrome, myasthenia gravis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, at screening, that requires use of immunosuppressives, glomerulonephritis, nephritic syndrome, Fanconi Syndrome or renal tubular acidosis within the past 2 years prior to the start of treatment. The following are exceptions to this criterion:

  1. Subjects with vitiligo or alopecia, hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement or psoriasis not requiring systemic treatment; patients with coeliac disease controlled by diet alone and patients without active disease in the last 5 years may be included after consultation with Chief Investigator.
  2. HBsAg carrier without active viral infection and under entecavir prophylaxis will be allowed.
* 7. History of (non-infectious) ILD/pneumonitis, current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
* 8. Active hepatitis B (HBV surface antigen [HBsAg] positive) or active hepatitis C. Virus testing is not essential for clinical trial feasibility assessment. Patients who have had or have resolved HBV infection or HCV infection in the past may participate in clinical trials. (Note: For HBsAg-, patient needs to be >6 months off antiviral treatment.)
* 9. Participants with past or resolved HBV infection are eligible only if they meet all of the following criteria*:

  1. Anti-HBc (+) (IgG or total Ig),
  2. HBV DNA undetectable,
  3. Absence of cirrhosis or fibrosis on prior imaging or biopsy,
  4. Absence of HCV co-infection or history of HCV co-infection.
  5. Access to a local Hepatitis B expert during and after the study. Such participants should be closely monitored for HBV reactivation. Consideration should be given to exclusion of all participants with HBV infection if comparator or combination study treatments are associated with a high risk of HBV infection reactivation are incompatible with anti-viral medications.
* 10. Known to have tested positive for human immunodeficiency virus (HIV) (positive HIV 1/2 antibodies) or active tuberculosis infection (clinical evaluation that may include clinical history, physical examination and radiographic findings, or tuberculosis testing in line with local practice). Active or prior documented history of primary immunodeficiency at screening. And HIV infection that is not well controlled. All of the following criteria are required to define an HIV infection that is well controlled:

  1. undetectable viral RNA,
  2. CD4+ count ≥350 cells/μL,
  3. no history of AIDS-defining opportunistic infection within the past 12 months, and stable for at least 4 weeks on the same anti-HIV medications (meaning there are no expected further changes in that time to the number or type of antiretroviral drugs in the regimen). If an HIV infection meets the above criteria, monitoring of viral RNA load and CD4+ count is recommended. Participants must be tested for HIV if acceptable by local regulations or an institutional IRB/IEC.
* 11. Patient with any of the following cardiac criteria:

  1. Mean QT interval corrected for heart rate (QTc) ≥ 470 ms calculated from electrogram (ECG) using Fridericia's correction
  2. Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG e.g. complete left bundle branch block, third degree heart block, second degree heart block, PR Interval >250 msec.
  3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, uncorrectable chronic hypokalemia, congenital long QT syndrome, family history (first-degree relatives) of long QT syndrome or unexplained sudden death under 40 years of age or concomitant medication known to prolong the QT interval
  4. Uncontrolled hypotension: systolic BP < 90 mmHg and/or diastolic BP 60 mmHg or clinically relevant orthostatic hypotension, including a fall in blood pressure of > 20 mmHg
  5. Atrial fibrillation with a ventricular rate >100 bpm on ECG at rest
  6. Symptomatic congestive heart failure (NYHA grade II-IV)
  7. Known reduced LVEF < 55%
  8. Prior or current cardiomyopathy of any etiology
  9. Prior or current acute myocardial infarction within the past 6 months
  10. Severe valvular heart disease
  11. Uncontrolled angina (Canadian Cardiovascular Society grade II-IV despite medical therapy)
  12. Stroke or transient ischaemic attack in prior to screening
  13. Acute coronary syndrome within 6 months prior to starting treatment
* 12. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 7 months after the last dose of Trastuzumab deruxtecan and Capecitabine or Rilvegostomig.
* 13. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
* 14. Current or prior use of immunosuppressive medication within 14 days before the first dose of investigational product is excluded. The following are exceptions to this criterion:

  1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intraarticular injection).
  2. Systemic corticosteroids at physiological doses not to exceed 10 mg/day of prednisone or equivalent.
  3. Steroids as premedication for hypersensitivity/infusion reactions and Receipt of live attenuated vaccine within 30 days prior to the first dose of study intervention. (Note: Participants should not receive live vaccine while receiving study intervention and up to 30 days after the last dose of study intervention.)
* 15. (For Rilvegostomig): Serious chronic gastrointestinal conditions associated with diarrhea (e.g., active inflammatory bowel disease); active non-infectious skin disease (including any grade rash, urticarial, dermatitis, ulceration, or psoriasis) requiring systemic treatment, active or prior documented autoimmune or inflammatory disorders requiring chronic treatment with steroids or other immunosuppressive treatment.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2028-10-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of AEs/SAEs | Through study completion, an average of 4 years
  To evaluate the safety and tolerability (by NCI-CTCAE v5.0)

SECONDARY OUTCOMES:
Pathologic CR(Pathological Complete Response) | Through study completion, an average of 1 year
  To assess by OP pathology review
EFS (Event-free survival) | Through study completion, an average of 4 years
  Modified Recist v1.1
OS (Overall survival) | Through study completion, an average of 4 years
  Kaplan-Meier method

CONTACTS AND LOCATIONS:
Overall Officials: Jeeyun Lee, Ph, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea